CLINICAL TRIAL: NCT02175511
Title: Cloud BP System Integrated With CPOE Improves Self-Management of the Hypertensive Patients: A Randomized Controlled Trial Study
Brief Title: A Randomized Controlled Trial for Hypertension Control by Integrating Cloud BP System and CPOE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NSC 100-2622-E-038-001-CC2
Record Dates: First submitted 2014-06-09; First posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Hypertension
Keywords: Home Blood Pressure; Computerized physician order entry (CPOE); Telemonitoring; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cloud-based home BP monitoring (Experimental): 170 were assigned to the experimental group
  Interventions: Device: Cloud-based home BP monitoring
- Traditional Care (No Intervention): 212 patients were assigned to the traditional care group (paper-based data)

INTERVENTIONS:
Device: Cloud-based home BP monitoring — a sphygmomanometer-style BP measurement device (Microlife®, "WatchBP Home") that stored and transmitted data to a secure cloud BP system directly via a General Packet Radio Service (GPRS) gateway through cell phone network.
  Arms: Cloud-based home BP monitoring

SUMMARY:
Importance: Less than fifty percent of patients with hypertensive disease manage to maintain their blood pressure (BP) within normal levels. Practical (Pragmatic) and sustainable models are needed in order to improve BP management in patients with hypertension.

Objective: To evaluate whether cloud BP system integrated with computerized physician order entry (CPOE) is useful for improving BP management as compared with traditional care.

DETAILED DESCRIPTION:
Design, Setting and Patients: A randomized clinical trial study of 382 adults recruited from 786 patients who had been diagnosed with hypertension and receiving treatment for hypertension in two district hospitals in the north of Taiwan. Physicians had access to cloud-based BP data from CPOE. Neither participants nor investigators were blinded to group assignment. The study was conducted for a period of seven months.

Interventions: Patients from two hospitals were randomized into a control group which received traditional care (n=212) and an intervention group (n=170) which received a cloud-based home BP monitoring device. The device measured and transmitted BP data to the cloud server, which was integrated with the CPOE system in the hospitals. Physicians could access the BP data during the patient encounter to adjust the antihypertensive therapy accordingly. Meanwhile, patients could browse their own BP data from their computers, smart phones, tablets and so on.

Primary Outcome(s) and Measure(s): The primary outcomes were control of systolic BP to less than 140 mm Hg and diastolic BP to less than 90 mm Hg at two, four and six months. The secondary outcomes were changes in BP and antihypertensive drug prescription at two, four and six months.

ELIGIBILITY:
Inclusion Criteria:

* Secondary hypertension
* Expectant mother
* Stroke, myocardial infarction or had surgery within 3 months
* Atrial fibrillation
* Inter-arm difference (IAD) >20 mm Hg
* Unsuitability as recognized by physicians.

Exclusion Criteria:

* Unable to participate in this trial for the whole process
* Lived alone and unable to read Text Message

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with controlled BP (<140/90 mm Hg) | Patients who participated in this trial will be followed for an expected average of 6 months

SECONDARY OUTCOMES:
The changes in BP and antihypertensive drug prescription | Patients who participated in this trial will be followed for an expected average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chuan Li, MD., PhD., Study Chair — Taipei Medical University; Peisan Lee, MA, Study Director — Taipei Medical University